CLINICAL TRIAL: NCT03922503
Title: Clinical Evaluation of Advanced Platelet Rich Fibrin With (DFDBA) Compared to Collagen Membrane With (DFDBA) in Treatment of Non-contained Intraosseous Defects in Stage III Periodontitis Patients: A Randomized Clinical Trial
Brief Title: Clinical Effect of APRF With DFDBA Compare to Collagen Membrane With DFDBA in Intraosseous Defect
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Najeeb Mohammed Mahyoub Ahmed, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01091495663
Record Dates: First submitted 2019-04-17; First posted 2019-04-22 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Intrabony Periodontal Defect
Keywords: Stage III periodontitis; APRF; Advanced Platelet Rich Fibrin; Demineralized freeze-dried bone allograft; DFDBA; Collagen Membrane; non-contained intraosseous defects; one wall intraosseous defects; combined 1- to 2-wall intraosseous defect
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Due to the type of intervention only the outcome assessor and the statistician will be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Advanced- platelets rich fibrin with DFDBA (Experimental): In A-PRF assigned group, one PRF will be cut into small pieces and added to the Demineralized freeze-dried bone allograft (DFDBA) in a ratio of 1:1 and the mixture is applied into the intraosseous defect, and the other will be used to prepare the membrane to cover the defect as a barrier. The mucoperiosteal flaps will be repositioned and secured in place using4-0 silk sutures.
  Interventions: Procedure: Advanced- platelets rich fibrin (A-PRF) with Demineralized freeze-dried bone allograft (DFDBA)
- Collagen membrane and DFDBA (Active Comparator): After debridement and intraoperative recordings, in the control group, Demineralized freeze-dried bone allograft (DFDBA) will be applied to the bone defect without overfilling and is protected by a collagen membrane, then interrupted sutures using 4-0 silk sutures will be placed to reposition the flaps.
  Interventions: Procedure: Collagen membrane with Demineralized freeze-dried bone allograft (DFDBA)

INTERVENTIONS:
Procedure: Advanced- platelets rich fibrin (A-PRF) with Demineralized freeze-dried bone allograft (DFDBA) — In A-PRF assigned group, one PRF will be cut into small pieces and added to the Demineralized freeze-dried bone allograft (DFDBA) in a ratio of 1:1 and the mixture is applied into the intraosseous defect, and the other will be used to prepare the membrane to cover the defect as a barrier.The mucoperiosteal flaps will be repositioned and secured in place using4-0 silk sutures.
  Arms: Advanced- platelets rich fibrin with DFDBA
Procedure: Collagen membrane with Demineralized freeze-dried bone allograft (DFDBA) — After debridement and intraoperative recordings, in the control group, Demineralized freeze-dried bone allograft (DFDBA) will be applied to the bone defect without overfilling and is protected by a collagen membrane, then interrupted sutures using 4-0 silk sutures will be placed to reposition the flaps.
  Arms: Collagen membrane and DFDBA

SUMMARY:
to assess the effectiveness of advanced PRF in combination of Demineralized freeze-dried bone allograft (DFDBA) as compared to collagen membrane in combination with Demineralized freeze-dried bone allograft (DFDBA) treatment of non-contained periodontal intraosseous defects in stage III periodontitis patients.

DETAILED DESCRIPTION:
Treatment of intraosseous periodontal defects represents a clinical challenge; these defects have been detected through clinical and radiographic examination in 18- 51 % of patients with periodontitis. They are often associated with persistent deep pockets and bleeding following conventional periodontal treatment. Complex regenerative periodontal therapy is advocated for management of these defects. The outcomes of regenerative periodontal therapy are positively correlated with the morphology of osseous defects. Non-contained defects are prevalent clinically and have been reported to have a low regenerative potential.

ELIGIBILITY:
Inclusion Criteria:

* Stage III periodontitis patient having at least one tooth with one wall or combined1- to 2-wall intraosseous defect ≥ 3 mm deep (assessed by trans-gingival probing, radiographic examination) with clinical attachment level (CAL) ≥ 5mm and pocket depth (PD) ≥ 6 mm.
* Defect not extending to a root furcation area
* Vital teeth
* Non-smokers.
* No history of intake of antibiotics or other medications affecting the periodontium in the previous 6 months.
* No periodontal therapy carried out in the past 6 months.
* Able to sign an informed consent form.
* Patients age between 25 and 50 years old.
* Patients who are cooperative, motivated, and hygiene conscious.
* Systemically free according to Cornell Medical Index

Exclusion Criteria:

* Pregnancy or breast feeding
* The presence of an orthodontic appliance
* Teeth mobility greater than grade I

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2019-09-30 (Actual); Primary Completion 2021-10-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in clinical attachment level (CAL) | CAL will be measured at base line, 3, 6, 9, 12 months postoperative
  CAL will be measured from the CEJ to the bottom of the gingival sulcus/periodontal pocket using UNC periodontal probe at six sites per tooth.

SECONDARY OUTCOMES:
Pobing Depth (PD) | PD will be measured at base line, 3, 6, 9, 12 months postoperative
  PD will be measured from the gingival margin to the bottom of the gingival sulcus/ periodontal pocket using UNC periodontal probe at six sites per tooth.
Gingival Recession Depth (RD) | RD will be measured at base line, 3, 6, 9, 12 months postoperative
  RD will be measured from the CEJ to the most apical extension of the gingival margin using UNC periodontal probe at six sites per tooth
Radiographic defect fill (IBD) | IBD will be measured at base line, 3, 6, 9, 12 months postoperative
  IBD will be measured from the alveolar bone crest to the base of the defect at baseline and after 6 months to detect the amount of bone fill Individually customized bite blocks and parallel-angle technique will be used to obtain standardized radiographs. Radiographs will be scanned and the radiographic IBD depth was measured by a computer-aided software program
Post-surgical patient satisfaction | After 12 months postoperative
  A 3-item questionnaire will be asked to the patients and shall use a 7-point answer scale These items will be: • Would you experience the same surgery another time?
  * Would you advice others with the surgery?
  * To what extent are you satisfied with the results?

CONTACTS AND LOCATIONS:
Overall Officials: Manal Hosny, Study Director — Cairo University
Locations (1):
- Faculty of dentistry cairo university, Cairo, Egypt

REFERENCES:
- [Result] Agarwal A, Gupta ND, Jain A. Platelet rich fibrin combined with decalcified freeze-dried bone allograft for the treatment of human intrabony periodontal defects: a randomized split mouth clinical trail. Acta Odontol Scand. 2016;74(1):36-43. doi: 10.3109/00016357.2015.1035672. Epub 2015 May 14. PMID 25972081
- [Result] Ainamo J, Bay I. Problems and proposals for recording gingivitis and plaque. Int Dent J. 1975 Dec;25(4):229-35. PMID 1058834
- [Derived] Almoliky N, Hosny M, Elbattawy W, Fawzy El-Sayed K. Low-Speed Platelet-Rich Fibrin Membrane in Conjunction With Demineralized Freeze-Dried Bone Allograft (DFDBA) Compared to Collagen Membrane With DFDBA in Noncontained Intraosseous Defects of Stage III Periodontitis: A Randomized Controlled Clinical Trial. Int J Dent. 2025 Feb 23;2025:6393105. doi: 10.1155/ijod/6393105. eCollection 2025. PMID 40028653